CLINICAL TRIAL: NCT02484469
Title: Educational Virtual Objects (The Virtual Human Project) Assessment Inserted in Learning Based on Team (Team-based Learning) in Leprosy Education on Undergraduate Medical Setting
Brief Title: Impact of the Virtual Human Project on Team-based Learning: A Randomized-controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Cristiane Comparin, Dr., Coordenação de Aperfeiçoamento de Pessoal de Nível Superior.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 001
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Leprosy
MeSH Terms: conditions — Leprosy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposed (Experimental): The Virtual Human Project videos and Team-Based learning session about leprosy
  Interventions: Device: The Virtual Human Project
- Unexposed (Placebo Comparator): Standard Team-Based learning session about leprosy

INTERVENTIONS:
Device: The Virtual Human Project — Virtual Human educational videos about leprosy
  Arms: Exposed

SUMMARY:
Team-based learning (TBL) is a learner-centered, instructor-directed strategy for small group active learning in large group educational settings. When TBL is conducted correctly, the students' performances are equivalent or improved in comparison to either lecture-based formats or more traditional small group learning models.1 Nevertheless, few studies have been published regarding the insertion of innovative audiovisual tools in the TBL context. The Virtual Human Project is described as powerful sequences of three dimension (3D) computer graphics video of the human body that aids learning by facilitating an understanding in relation to a specific subject. The Virtual Human is composed by video sequences combining anatomy, physiology, and morphology in the context of various diseases. There are video sequences available for many disciplines, including dermatology and with capacity to produce anatomical structures by 3D printer. Despite the incredible potential applications of the Virtual Human, few studies have assessed its impact on medical education. The investigators did not find any study evaluating TBL with the insertion of iconographic educational material that assessed whether this intervention could change the learning progress of students. This is the aim of the present study, by comparing students tests scores after a TBL session with the VIrtual Human videos about leprosy or a standard TBL session, and to evaluate the student's satisfaction with the Virtual Human videos.

ELIGIBILITY:
Inclusion Criteria:

* undergraduate medical students in the third year of Medical School at the Federal University of Mato Grosso do Sul.

Exclusion Criteria:

* students previously exposed to dermatologic research, extracurricular activities involving dermatology or dermatology rotation in that year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Average of Individual readiness assessment test (IRAT) grades | One year
  The average of the IRAT scores achieved by students

SECONDARY OUTCOMES:
The Average of group readiness assessment test (GRAT) grades | One year
  The average of the GRAT scores achieved by students
The Average of clinical case scores | One year
  The average of the clinical case scores achieved by students